CLINICAL TRIAL: NCT01160003
Title: A Randomised, Double-blind, Placebo-controlled, Dose Ascending,3-way Crossover Study to Assess the Pharmacokinetics, Safety Andtolerability of Repeat Inhaled Doses of Nebulised GW870086X Inhealthy Adult Male Volunteers.
Brief Title: A Blinded, Dose Ascending Study to Assess the Pharmacokinetics, Safety and Tollerability of Repeat Inhaled Doses of Nebulised GW870086X in Healthy Adult Male Volunteers.
Acronym: SIG
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 113209
Record Dates: First submitted 2010-07-08; First posted 2010-07-12 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Asthma
Keywords: ACTH stimulation test; Pharmacokinetics; Nebules; Cortisol
MeSH Terms: conditions — Asthma | interventions — GW870086X

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Period 1 (Experimental): 5mg of GW870086X or placebo will be given once daily for 14 days.
  Interventions: Drug: GW870086X; Drug: Placebo
- Treatment Period 2 (Experimental): GW870086X (5mg or 8.75mg) or placebo will be given once daily for 14 days. In a randomised dose escalating manor following on from treatment period 1.
  Interventions: Drug: GW870086X; Drug: Placebo
- Treatment Period 3 (Experimental): 8.75mg of GW870086X or placebo will be given once daily for 14 days.
  Interventions: Drug: GW870086X; Drug: Placebo

INTERVENTIONS:
Drug: GW870086X — 5mg and 8.75mg GW870086X once daily for 14 days in separate traetment periods.
Drug: Placebo — placebo will be randomly inserted into one of the treatment periods following the treatment sequences outlined in the protocol.

SUMMARY:
This study is a randomised, double-blind, placebo-controlled, dose ascending, 3-way crossover study in healthy adult male volunteers. The primary objective of the study is to assess the pharmacokinetics of 14 days dosing of GW870086X administered via nebules formulation. The secondary objective is to assess the safety and tolerability of repeat doses of nebulised GW870086X.

DETAILED DESCRIPTION:
GW870086X is a potent glucocorticoid agonist in human in vitro functional assays that is under development as an inhaled treatment for asthma in children. This study will determine the PK characteristics and assess the safety and tolerability of the nebules formulation of GW870086X in healthy volunteers after 14 days of dosing.

This is the first clinical study that will be assessing the nebules formulation. The purpose of this study is to ensure that the doses that have been selected have a good safety profile in line with what has been found in the previous DPI formulation studies, and to assess the PK profile after single (Day 1) and repeat dose (Day 14) to select appropriate doses for future studies with the nebules formulation. This study will also provide additional safety cover with the nebules formulation given over a longer duration than studied previously with the DPI formulation before moving into the paediatric programme. This study is designed to give at least 5-fold cover for the highest dose to be studied in future paediatric programmes. During this study cortisol production will be assessed by measuring 24 hour cortisol profile in serum and urine as well as performing an ACTH stimulation test. Two doses (5mg and 8.75mg) have been selected. These doses are 5 and 10 times higher than the anticipated maximum clinical dose. The doses have been selected to ensure sufficient safety cover in future paediatric studies as well as to confirm the absence of significant adrenal inhibition at doses that would be expected to cause complete inhibition of cortisol production with traditional steroids.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria apply:

  1. Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
  2. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
  3. AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
  4. Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 90-95 hours post-last dose.
  5. Body weight, men ≥ 50 kg and BMI within the range 19.0 - 29.0 kg/m2 (inclusive).
  6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
  7. Single QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

  1. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
  2. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
  3. A positive pre-study drug/alcohol screen.
  4. A positive test for HIV antibody.
  5. History of regular alcohol consumption within 6 months of the study defined as:

     For EU sites: an average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.
  6. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
  7. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
  8. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
  9. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
  10. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
  11. Unwillingness or inability to follow the procedures outlined in the protocol.
  12. Subject is mentally or legally incapacitated.
  13. Subjects who are kept due to regulatory or juridical order in an institution.
  14. Subjects who are in military service.
  15. History of sensitivity to heparin or heparin-induced thrombocytopenia.
  16. Subjects who have asthma or a history of asthma.
  17. Subject is a smoker or an ex-smoker with a smoking history of > 5 pack years (Pack years = (cigarettes per day smoked/20) x number of years smoked)).
  18. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-07-29 (Actual); Primary Completion 2010-11-05 (Actual); Study Completion 2010-11-05 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of GW870086X and GW870086X pharmacokinetic parameters (including AUC, Cmax, t1/2 and tmax) | 3 months

SECONDARY OUTCOMES:
Adverse Events | 3 months
Clinically relevant changes in safety parameters:Clinical laboratory tests (clinical chemistry, haematology, urinalysis), 12-Lead ECG data; including QT, QTc, HR, QRS and RR intervals, Vital signs: systolic and diastolic blood pressure, pulse rate | 3 months
Serum cortisol weighted mean over 24 hours | 3 months
Urine cortisol excretion over 24 hours | 3 months
ACTH stimulation test (Period 3 only) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 113209 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/113209?search=study&search_terms=113209#rs
- Available data/document: Annotated Case Report Form: 113209 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 113209 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113209 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113209 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113209 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113209 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113209 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register